CLINICAL TRIAL: NCT03064789
Title: Estudio epidemiológico de la evolución clínica y microbiológica en Pacientes Tratadas Por un Episodio Agudo de Candidiasis Vulvovaginal
Brief Title: Epidemiological Study in Subjects With Vulvovaginal Candidiases
Status: Completed | Type: Observational
Sponsor: Dr. Santiago Palacios (Other)
Responsible Party: Sponsor-Investigator, Dr. Santiago Palacios, MD - Gynecologyst, Instituto Palacios
Organization: Instituto Palacios (Other)
Other Study IDs: IP-01-2016
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Vulvovaginal Candidiases
Keywords: Candidiases; Vaginal Infections
MeSH Terms: conditions — Candidiasis; Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with candidiases infection: Women that are prescribed treatment with clotrimazole: 500 mg. and probiotics (routine clinical practice)

SUMMARY:
Epidemiological study about the clinical and microbiological progress in subjects under treatment for a severe vulvovaginal candidiases episody

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women between 18 and 50 years of age at time of screening
* With diagnosis and symptomatology of VVC

Exclusion Criteria:

* Pregnant women
* Diabetes Mellitus
* Women witihin three months after a delivery or misbirth
* Women with vaginal or genital infection symptomatology other than candidiases that needs antibiotic treatment
* Vaginal probiotics use within last three months
* Undiagnosed abnormal genital hemorrhage

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with VVC symptomatology and positive culture
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Estimate cure rate in women with severe vuvovaginal candidiases infection | At 3 months
  Women must require antimicotic treatment plus vaginal probiotic following the habitual therapeutic standards

SECONDARY OUTCOMES:
Estimate recurrences | At 6 months
  It will be consider recurrences an asymptomatic period for 7-10 days and a negative culture
Estimate recurrences | At 12 months
  It will be consider recurrences an asymptomatic period for 7-10 days and a negative culture
Evaluate the link between symptomatology and negative culture | At 3 months
Evaluate the effectiveness of probiotic treatment by physician | At 3 months
  A gynecological exploration will be performed
Evaluate the effectiveness of probiotic treatment by patient. A satisfaction questionnaire will be performed | At 3 months
  The subject will be asked how long the symptoms lasted and the gravity of them

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, PI, Principal Investigator — Instituto Palacios
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No